CLINICAL TRIAL: NCT01020032
Title: Effect of Music Therapy on Chronic Pain in Hospitalized Patients in a Pain Center
Brief Title: Effect of Music Therapy on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Musicothérapie Applications et Recherches Cliniques (Other)
Collaborators: Centre d'Evaluation et du Traitement de la Douleur CHU Saint-Eloi (Unknown); Unité de Recherche Clinique et Epidémiologie (DIM) CHU Arnaud de Villeneuve (Unknown); Centre Mémoire de Ressource et de Recherche équipe INSERM U888 CHU Montpellier (Unknown)
Responsible Party: GUETIN, AMARC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMARC 200801
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Pain
Keywords: Music therapy; Pain; Anxiety; Depression; Controlled randomized trial
MeSH Terms: conditions — Chronic Pain; Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Music therapy (Experimental): Individual receptive music therapy by "U sequence" method
  Interventions: Other: Individual receptive music therapy by "U sequence" method

INTERVENTIONS:
Other: Individual receptive music therapy by "U sequence" method — During the hospitalization, the intervention group benefited from at least 2 daily sessions of music therapy between day 0 and day 10, and continued the musicotherapy at home until day 60.

SUMMARY:
The aim of study is to assess the effects of this new music therapy technique on pain treatment, anxiety and depression and on medicinal consumption.

DETAILED DESCRIPTION:
The "U" technique is a music therapy method of recent use developed by taking into account recommendations of the scientific literature. The objective of the study is to evaluate this method on chronic painful patients presenting a lumbago, a fibromyalgia, an inflammatory or neurological pathology. During the hospitalization, the intervention group benefited from at least 2 daily sessions of music therapy between day 0 and day 10, and continued the musicotherapy at home until day 60. The evaluated criteria are pain, depression and anxiety and their evolution after 60 days of treatment (since the inclusion). The evaluation at day 90 allows to test the persistence of the effect of the music therapy 90 days later.

ELIGIBILITY:
Inclusion Criteria:

* Have a pain for more than 6 months
* Pain of neurological origin (fibromyalgia, algodystrophies), or skeletal musculous (back, sciatic nerve)
* Speak and read French fluently
* Wrote consent of patients
* Benefit from the standard treatment : Intravenous treatment (tranquillizer, antidepressive) the first 5 days, 2 time by day (in the morning and evening), followed by the intermediary orally up to the exit (prescribed doses and at request)

Exclusion Criteria:

* Time of hospitalization < 8 days
* Reflex epilepsy history
* Major insufficiency of auditory function
* Patient with a strong possibility of not compliance to the protocol or of abandon in the course of study
* Presence of an illness threatening vital forecast during period envisaged for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Score on a Visual Analogical Scale (VAS) for actual pain | Day 0, day 5, day 10, day 60 and day 90

SECONDARY OUTCOMES:
Score on the Hospital Anxiety and Depression (HAD) Scale | Day 0, day 5, day 10, day 60 and day 90
Medicinal consumption | Before hospitalization, day 0, day 5, day 10, day 60 and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane GUETIN, PhD, Principal Investigator — Association de Musicothérapie Applications et Recherches Cliniques
Locations (1):
- CHRU Saint Eloi, Centre d'Evaluation et du Traitement de la Douleur, Montpellier, France

REFERENCES:
- [Background] Roy M, Peretz I, Rainville P. Emotional valence contributes to music-induced analgesia. Pain. 2008 Jan;134(1-2):140-7. doi: 10.1016/j.pain.2007.04.003. Epub 2007 May 25. PMID 17532141
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Guetin S, Portet F, Picot MC, Pommie C, Messaoudi M, Djabelkir L, Olsen AL, Cano MM, Lecourt E, Touchon J. Effect of music therapy on anxiety and depression in patients with Alzheimer's type dementia: randomised, controlled study. Dement Geriatr Cogn Disord. 2009;28(1):36-46. doi: 10.1159/000229024. Epub 2009 Jul 23. PMID 19628939
- See also: AMARC association is specialized in applications and clinical researches in music therapy — http://www.amarc.fr